CLINICAL TRIAL: NCT00958815
Title: Human Atherosclerotic Plaque Inflammation Imaged Using PDG-PET/CT
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kevin Yarasheski, Professor of Medicine, Cell Biology & Physiology, Physical Therapy, Washington University School of Medicine
Other Study IDs: 18FDG (completed); DK-020579
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Insulin Resistance; Atherosclerosis; Cardiovascular Disease; HIV/AIDS; HIV Infections
Keywords: vascular imaging; diabetes; rupture prone plaques; HIV; treatment experienced
MeSH Terms: conditions — Insulin Resistance; Atherosclerosis; Cardiovascular Diseases; Acquired Immunodeficiency Syndrome; HIV Infections; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV-seronegative with no CVD risk factors: Healthy, 35-60 yr old HIV-seronegative men and women with no CVD risk factors (normal fasting glucose tolerance, normal fasting lipid/lipoprotein levels, normotensive, waist circumference <102cm (men) and <88cm (women).
- HIV+ with CVD risk factors: 35-60 yr old HIV-infected men and women with insulin resistance, dyslipidemia, hypertension, and central adiposity.

SUMMARY:
People with diabetes are at increased risk for atherosclerosis and have high CVD morbidity and mortality rates. Tools for detecting and quantifying atherosclerotic pro/regression in people with diabetes and other CVD risk factors lack sensitivity and specificity for molecular level events that occur during the early stages of atherogenesis. Inflammatory macrophage infiltration in the vessel endothelium is an early, molecular level proatherogenic event. Activated macrophages consume glucose at a high rate. Novel in vivo radiotracer PET/CT techniques have been developed to detect, image and quantify molecular level events like macrophage inflammation and glucose utilization (18FDG) in human vessels. We propose to develop and test this novel technique in the Center for Clinical Imaging Research (CCIR) at WUMS. We propose that HIV-infected people with significant CVD risk profiles are a suitable, unique human model for testing these novel imaging techniques. HIV-infected people taking anti-HIV medications develop insulin resistance, T2DM, dyslipidemia, central adiposity, and hypertension. HIV replicates in macrophages and represents a chronic proinflammatory condition. Recent data indicate that HIV+ CVD risk have greater risk for atherosclerosis and MI than HIV-negative people. To test feasibility, we hypothesize that: a.18FDG-PET/CT imaging will detect more macrophage glucose uptake and inflammation in the carotid and aorta arteries of HIV-infected people with CVD risk than in HIV-negative controls; b. radiotracer PET/CT measures of proatherogenic processes will correlate with carotid intima media thickness; a standard measure of carotid atherosclerotic burden. We propose to obtain pilot data that shows feasibility for a novel analytical approach that will expand capabilities for researchers interested in studying the links between diabetes, inflammation, and CVD in humans.

ELIGIBILITY:
Inclusion Criteria for HIV+ group:

* confirmed HIV+ status
* 35-60 years old
* stable ART for at least the past 4 mos
* CD4 count >200 cells/µL
* HIV RNA <40copies/mL
* fasting glucose=100-126 mg/dL
* 2hr-oGTT glucose=140-200mg/dL
* fasting triglycerides >150mg/dL
* HDL-cholesterol <40mg/dL (men), <50mg/dL (women)
* resting blood pressure>130/85mmHg
* waist circumference >102cm(men), >88cm(women)
* BMI 25-35 kg/m2

For HIV-negative control group:

* Confirmed HIV negative status
* 35-60 years old
* fasting glucose<100mg/dL,
* 2hr-oGTT glucose<140mg/dL
* fasting triglycerides<150mg/dL
* HDL-cholesterol >40mg/dL (men), >50mg/dL(women)
* normal BP (<130/85mmHg)
* no central adiposity (waist circ.<102cm(men), <88cm(women)
* BMI (25-35 kg/m2)

Exclusion Criteria for both groups:

* history of heart disease, MI, stroke, transient ischemic attack, kidney or liver disease (active hepatitis B or C), dementia
* statins, fibrates, TZDs, antihypertensives, low dose aspirin, or other prescribed/over-the-counter agents with anti-inflammatory properties
* cocaine and methamphetamine users
* serum creatinine >1.5 mg/dL
* pregnant women
* cognitive impairment that limits ability to provide voluntary informed consent

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited through the AIDS Clinical Trials Unit (ACTU), Washington University Infectious Diseases Clinics, primary care physicians in the community who refer patients to these clinics and Volunteers for Health (VFH).
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Standard uptake values (SUV) for 18Fluoro-deoxyglucose in the carotid vessels and aorta of HIV-infected people with cardiovascular disease risk factors and compared to the same in HIV-seronegative people with no cardiovascular disease risk factors. | Baseline

SECONDARY OUTCOMES:
Carotid intima media thickness measures will be compared to carotid 18FDG SUV. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kevin E Yarasheski, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Yarasheski KE, Laciny E, Overton ET, Reeds DN, Harrod M, Baldwin S, Davila-Roman VG. 18FDG PET-CT imaging detects arterial inflammation and early atherosclerosis in HIV-infected adults with cardiovascular disease risk factors. J Inflamm (Lond). 2012 Jun 22;9(1):26. doi: 10.1186/1476-9255-9-26. PMID 22726233
- See also: Publication — http://www.journal-inflammation.com/content/9/1/26/abstract